CLINICAL TRIAL: NCT04480918
Title: University of Iowa Interventional Psychiatry Service Patient Registry
Status: Recruiting | Type: Observational
Sponsor: Mark Niciu (Other)
Responsible Party: Sponsor-Investigator, Mark Niciu, Assistant Professor, University of Iowa
Organization: University of Iowa (Other)
Other Study IDs: 202003055
Record Dates: First submitted 2020-07-02; First posted 2020-07-22 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2024-08

CONDITIONS: Treatment Resistant Depression; Major Depressive Episode; Major Depression; Major Depressive Disorder; Bipolar Disorder; Bipolar Depression; Obsessive-Compulsive Disorder
Keywords: Electroconvulsive Therapy; Transcranial Magnetic Stimulation; Ketamine; Esketamine
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Depressive Disorder, Major; Bipolar Disorder; Obsessive-Compulsive Disorder | interventions — Transcranial Magnetic Stimulation; Ketamine; Esketamine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Biospecimen Retention: Samples With DNA — blood, saliva and cheek swabs for epi/genetic expression
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Major Depressive Episode: After referral to the University of Iowa's Interventional Psychiatry Clinic, the patient will be clinically evaluated and, if appropriate, commence the procedural-based treatment course.
  Interventions: Device: Electroconvulsive Therapy (ECT); Device: Transcranial Magnetic Stimulation (TMS); Drug: Ketamine; Drug: Esketamine; Device: Deep Transcranial Magnetic Stimulation (dTMS)

INTERVENTIONS:
Device: Electroconvulsive Therapy (ECT) — ECT for the treatment of treatment-resistant depression OR Bipolar Disorder in an active major depressive episode
Device: Transcranial Magnetic Stimulation (TMS) — TMS for the treatment of treatment-resistant depression in an active major depressive episode
Drug: Ketamine — Intravenous ketamine infusion for the treatment of treatment-resistant depression in an active major depressive episode
Drug: Esketamine — Intranasal esketamine insufflation for the treatment of treatment-resistant depression in an active major depressive episode
Device: Deep Transcranial Magnetic Stimulation (dTMS) — TMS for the treatment of OCD

SUMMARY:
The purpose of this study is to examine the effects of interventional/procedural therapies for treatment-resistant depression (TRD) and Obsessive-Compulsive Disorder (OCD). These treatments include electroconvulsive therapy (ECT), transcranial magnetic stimulation (TMS), racemic ketamine infusion and intranasal esketamine insufflation. The investigators will obtain various indicators, or biomarkers, of a depressed individuals' state before, during, and/or after these treatments. Such biomarkers include neurobehavioral testing, neuroimaging, electroencephalography, cognitive testing, vocal recordings, epi/genetic testing, and autonomic nervous system measures (i.e. "fight-or-flight" response). The results obtained from this study may provide novel antidepressant treatment response biomarkers, with the future goal of targeting a given treatment to an individual patient ("personalized medicine").

DETAILED DESCRIPTION:
Treatment response biomarkers in TRD and OCD have been and will remain an active area of research. Interventional treatments in psychiatry, e.g. ECT, TMS, racemic ketamine infusions and intranasal esketamine insufflations, offer exciting opportunities for biomarker discovery due their procedural nature (obviating concerns for treatment non-adherence in non-supervised settings), more rapid-onset, and larger effect sizes than typically seen with traditional antidepressant medications or evidence-based psychotherapies. Although no well-replicated TRD biomarkers have been approved for standard clinical use, several potential biomarkers have been investigated across multiple modalities, i.e. neuroimaging(1,2), autonomic function(3,4), genetics(5-7), electroencephalography (EEG) (8,9), and computational analysis of behavior or speech(10). These studies have promising early results but often insufficient predictive power at the subject-level. The investigators anticipate that combinatorial, multimodal biomarkers will enhance predictive power and, as a result, improve treatment personalization in major depression.

The University of Iowa Interventional Psychiatry Service Patient Registry systematically collects data from TRD and OCD patients undergoing procedural treatment(s) for major depression. First, the investigators seek to replicate and/or extend discoveries from prior investigations, e.g. TMS-induced autonomic changes as positive predictors of antidepressant efficacy. The investigators will also compare and contrast differences, not only in response to a given therapy, but also how individual subjects respond across different treatment modalities, e.g. how does functional connectivity in the brain change in response to an effective course of TMS as opposed to ECT? Such findings could inform the future development of clinical guidelines; this is especially critical as some of these treatment modalities have only recently been approved for TRD by the U.S. Food and Drug Administration, e.g. intermittent theta burst stimulation (iTBS) and intranasal esketamine insufflation and dTMS for OCD.

Next, a longitudinal database may also be valuable for future biomarker discovery and/or replication in independent samples, i.e. an epigenetic signature of antidepressant treatment response to an interventional modality identified by another research group. Similarly, this patient registry could be valuable for collaborative research with other institutions administering interventional treatments in psychiatry.

ELIGIBILITY:
INCLUSION CRITERIA:

1. 18-99 years of age
2. English-speaker with a level of understanding sufficient to agree to clinical treatment with a treatment modality offered by the Interventional Psychiatry Service, all required research procedures, and sign an informed consent document
3. Clinical diagnosis of a major depressive episode in the context of major depressive disorder or bipolar disorder or treatment-resistant OCD evaluated by a provider on the Interventional Psychiatry Service and felt to be an appropriate candidate for clinical treatment with a treatment modality offered by the Interventional Psychiatry Service.

EXCLUSION CRITERIA:

1. Age less than 18 years
2. A primary neuropsychiatric diagnosis that is not either major depressive disorder or bipolar disorder
3. Serious, unstable medical conditions/problems including hepatic, renal, gastroenterologic, respiratory, cardiovascular, endocrinologic, neurologic, immunologic, or hematologic disease, e.g. uncontrolled asthma, uncontrolled hyper/hypothyroidism or active cancer.
4. Involuntary commitment to psychiatry inpatient units
5. If patients have one or more of the following MRI Exclusion criteria, they will not be able to participate in those aspects of this study:

   1. The presence of an implanted device including pacemaker, coronary stent, defibrillator, or neurostimulation device that is not MRI-compatible
   2. The presence of ferromagnetic objects in the body, i.e. bullets, shrapnel, and/or metal slivers
   3. Clinically-significant claustrophobia
   4. Clinically-significant hearing loss
   5. Pregnant or nursing women or women of child bearing potential not using at least one medically accepted means of contraception (to include oral, injectable, or implant birth control, condom or diaphragm with spermicide, intrauterine devices (IUD), tubal ligation, abstinence, or partner with vasectomy)
   6. The presence of any medical illness likely to alter brain morphology and/or physiology (e.g., hypertension, diabetes) even if controlled by medications

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (18-99 years old) in a current major depressive episode in the context of major depressive disorder (MDD) or bipolar disorder (BD) will be recruited for this protocol. Adult patients received TMS for OCD will also be recruited. All treatment will be in addition to the patient's clinical care with the University of Iowa's Interventional Psychiatry Service for treatment-resistant major depression or OCD, and the decision to participate, withdraw from participation or not participate will if not affect clinical care decision-making. We appreciate that minority groups tend to be underrepresented in neuropsychiatric research studies. Therefore, we will make a concerted effort to keep the proportion of racial/ethnic minorities recruited consistent with the demographics of the surrounding communities.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-11-02 (Actual); Primary Completion 2050-08 (Estimated); Study Completion 2050-08 (Estimated)

PRIMARY OUTCOMES:
Montgomery-Åsberg Depression Rating Scale (MADRS) Pre-Post Change | Pre-assessment will be obtained within approximately 1 week of starting treatment. Post-assessment will be obtained as close as possible following completion of treatment course (usually 4-6 weeks later).
  For patients with TRD, the MADRS will be administered. The MADRS contains 10 items, and each item is scored 0-6. These item scores are summed to create a scale score; thus, scale scores range from 0 to 60. A scale score of 0 indicates the absence of depressive symptoms, while a score of 60 indicates severe depression. The primary outcome is the mean change in total MADRS score. A decrease in the mean MADRS score indicates a decrease (or improvement) in depressive symptoms, whereas an increase in the mean MADRS score indicates an increase (or worsening) in depressive symptoms.
Yale-Brown Obsessive Compulsive Scale | Pre-assessment will be obtained within approximately 1 week of starting treatment. Post-assessment will be obtained as close as possible following completion of treatment course (usually 4-6 weeks later).
  For patients with OCD, the YBOCS will be administered. Questions on the YBOCS examine the amount of time spent thinking and acting on obsessions and compulsions, how much impairment or distress is caused, and how much resistance and control the participant has over their thoughts or behavior.

SECONDARY OUTCOMES:
Clinical Global Impression/Severity (CGI) Pre-Post Change | Pre-assessment will be obtained within approximately 1 week of starting treatment. Post-assessment will be obtained as close as possible following completion of treatment course (usually 4-6 weeks later).
  The CGI is a clinician-measured scale of 3 items: Severity of Illness (item 1), Global Improvement (item 2), and Efficacy Index (item 3). Items 1 and 2 are rated on a 7-point Likert scale (1=normal, 7=among the most extremely ill patients) with a possible response of "not assessed." Item 3 is rated on a 4-point Likert scale from "none" to "outweighs therapeutic effect." Items 1 and 3 are assessed in relation to last clinical encounter (if possible).
Generalized Anxiety Disorder, 7-item (GAD-7) Pre-Post Change | Pre-assessment will be obtained within approximately 1 week of starting treatment. Post-assessment will be obtained as close as possible following completion of treatment course (usually 4-6 weeks later).
  The GAD-7 is the self-reported anxiety questionnaire which scores each of the 7 symptoms of Generalized Anxiety Disorder in the last two weeks on a 4-point scale, i.e. 0 ("not at all"), 1 ("several days"), 2 ("over half the days") and 3 ("nearly every day"). Functional impairment is also assessed from "Not difficult at all" to "Extremely difficult."
Montreal Cognitive Assessment (MoCA) Pre-Post Change | Pre-assessment will be obtained within approximately 1 week of starting treatment. Post-assessment will be obtained as close as possible following completion of treatment course (usually 4-6 weeks later).
  The MoCA is a 30-point screening instrument for detecting cognitive dysfunction. It is used to assess the following cognitive domains: visuospatial/executive, naming, memory, attention, language, abstraction, delayed (short-term memory recall), and orientation.
Patient Health Questionnaire, 9-item (PHQ-9) Pre-Post Change | Pre-assessment will be obtained within approximately 1 week of starting treatment. Post-assessment will be obtained as close as possible following completion of treatment course (usually 4-6 weeks later).
  The PHQ-9 is the self-reported depression module of the PHQ, which scores each of the 9 symptoms of a major depressive episode on a 4-point scale, i.e. 0 ("not at all"), 1 ("several days"), 2 ("more than half the days") and 3 ("nearly every day"). Functional impairment is also assessed from "Not difficult at all" to "Extremely difficult."
Temperament and Character Inventory (TCI) Pre-Post Change | Pre-assessment will be obtained within approximately 1 week of starting treatment. Post-assessment will be obtained as close as possible following completion of treatment course (usually 4-6 weeks later).
  The TCI is a 240-item questionnaire. It operates with seven dimensions of personality traits, i.e. four so-called temperaments: Novelty Seeking (NS), Harm Avoidance (HA), Reward Dependence (RD), and Persistence (PS), and three so-called characters: Self-Directedness (SD), Cooperativeness (CO) and Self-Transcendence (ST). Each of these traits has a varying number of subscales.

OTHER OUTCOMES:
Actigraphy Pre-Post Change | Pre-assessment will be obtained within approximately 1 week of starting treatment. Post-assessment will be obtained as close as possible following completion of treatment course (usually 4-6 weeks later).
  The patient will be asked to continuously wear a Fitbit wristband to monitor gross motor activity, e.g. foot steps. Changes in gross motor activity throughout the day will also provide data on circadian rhythmicity (sleep-wake cycles).
Candidate Gene (DNA) Polymorphisms | The genetic specimen will be obtained within approximately 1 week of starting treatment (likely with the baseline epigenetic sample.
  The investigators will obtain tissue samples, e.g. blood, saliva, and/or cheek swabs, and DNA will be isolated and extracted. Data on genetic polymorphisms (differences) that have been demonstrated or hypothesized to play a functional role in major depression, e.g. the brain derived neurotrophic factor (BDNF) rs6265 (val66met) single nucleotide polymorphism, will be obtained. These genotypes (genetic data) will then be correlated with antidepressant response.
Electroencephalography (EEG) Pre-Post Change | Pre-assessment will be obtained within approximately 1 week of starting treatment. Post-assessment will be obtained as close as possible following completion of treatment course (usually 4-6 weeks later).
  The investigators will obtain task-free ("resting state") rs-EEG [detecting electrical signals in the brain] at baseline and in response to interventional treatments for treatment-resistant depression.
Epigenetic (Experience-Based) DNA Modifications Pre-Post Change | The initial specimen will be obtained within approximately 1 week of starting treatment. The post-specimen will be obtained as close as possible following completion of treatment course (usually 4-6 weeks later).
  The investigators will obtain tissue samples, e.g. blood, saliva, and/or cheek swabs, at baseline and in response to interventional treatments for treatment-resistant depression. DNA will be isolated and extracted. Data on epigenetic (experience-based) modifications to the DNA that have been demonstrated or hypothesized to play a functional role in major depression, e.g. global methylation changes, will be obtained. Changes in epigenetic status, e.g. global DNA methylation changes pre- and post-treatment, will then be correlated with antidepressant response.
Facial Expression Analysis Pre-Post Change | Pre-assessment will be obtained within approximately 1 week of starting treatment. Post-assessment will be obtained as close as possible following completion of treatment course (usually 4-6 weeks later).
  Facial recognition software, FaceX (FaceX LLC) will be used to record and analysis facial features at rest and evoked by interview questions and emotionally provocative videos.
Galvanic Skin Response Pre-Post Change | Pre-assessment will be obtained within approximately 1 week of starting treatment. Post-assessment will be obtained as close as possible following completion of treatment course (usually 4-6 weeks later).
  Galvanic skin response as a surrogate marker of autonomic reactivity will be obtained in response to the presentation of emotional stories or images.
Heart Rate Variability Pre-Post Change | Pre-assessment will be obtained within approximately 1 week of starting treatment. Post-assessment will be obtained as close as possible following completion of treatment course (usually 4-6 weeks later).
  Heart rate variability as a surrogate marker of autonomic reactivity will be obtained in response to the presentation of emotional stories or images.
National Institutes of Health (NIH) Toolbox(R) Pre-Post Change | Pre-assessment will be obtained within approximately 1 week of starting treatment. Post-assessment will be obtained as close as possible following completion of treatment course (usually 4-6 weeks later).
  The NIH Toolbox is a comprehensive set of neurobehavioral assessments that assess multiple neuropsychiatric domains. We will perform the cognitive and emotional batteries in this study.
Pupillometry Pre-Post Change | Pre-assessment will be obtained within approximately 1 week of starting treatment. Post-assessment will be obtained as close as possible following completion of treatment course (usually 4-6 weeks later).
  Pupillometry (pupil diameter measurements) as a surrogate marker of autonomic reactivity will be obtained in response to the presentation of emotional stories or images.
Resting State Functional Magnetic Resonance Imaging (rs-fMRI) Pre-Post Change | The initial imaging session will be obtained within approximately 1 week of starting treatment. The post-treatment imaging session occur as close as possible following completion of treatment course (usually 4-6 weeks later).
  The investigators will obtain task-free ("resting state") rs-fMRI [detecting blood oxygen-level dependent (BOLD) signal in the brain] at baseline and in response to interventional treatments for treatment-resistant depression.
Structural Magnetic Resonance Imaging (MRI) Pre-Post Change | The initial imaging session will be obtained within approximately 1 week of starting treatment. The post-treatment imaging session occur as close as possible following completion of treatment course (usually 4-6 weeks later).
  The investigators will obtain structural brain imaging at baseline and in response to interventional treatments for treatment-resistant depression.
Vocal Pattern Detection Pre, During and Post-Change | Pre-assessment will be obtained within approximately 1 week of starting treatment. Interim assessments will occur weekly during treatment. Post-assessment will be obtained as close as possible following completion of treatment course.
  The patient will be asked to read standardized passages, i.e. Grandfather Passage and Rainbow Passage, and answer questions about daily life and interests while being recorded. These recordings will be transcribed and analyzed for vocal tone, inflection, word choice, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Mark J Niciu, M.D., Ph. D., Principal Investigator — University of Iowa Hospitals & Clinics; Nicholas T Trapp, M.D., M.S., Principal Investigator — University of Iowa Hospitals & Clinics
Locations (1):
- University of Iowa Health Care, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Levy A, Taib S, Arbus C, Peran P, Sauvaget A, Schmitt L, Yrondi A. Neuroimaging Biomarkers at Baseline Predict Electroconvulsive Therapy Overall Clinical Response in Depression: A Systematic Review. J ECT. 2019 Jun;35(2):77-83. doi: 10.1097/YCT.0000000000000570. PMID 30628993
- [Background] Cash RFH, Cocchi L, Anderson R, Rogachov A, Kucyi A, Barnett AJ, Zalesky A, Fitzgerald PB. A multivariate neuroimaging biomarker of individual outcome to transcranial magnetic stimulation in depression. Hum Brain Mapp. 2019 Nov 1;40(16):4618-4629. doi: 10.1002/hbm.24725. Epub 2019 Jul 22. PMID 31332903
- [Background] Iseger TA, Padberg F, Kenemans JL, Gevirtz R, Arns M. Neuro-Cardiac-Guided TMS (NCG-TMS): Probing DLPFC-sgACC-vagus nerve connectivity using heart rate - First results. Brain Stimul. 2017 Sep-Oct;10(5):1006-1008. doi: 10.1016/j.brs.2017.05.002. Epub 2017 May 12. PMID 28545770
- [Background] Cabrerizo M, Cabrera A, Perez JO, de la Rua J, Rojas N, Zhou Q, Pinzon-Ardila A, Gonzalez-Arias SM, Adjouadi M. Induced effects of transcranial magnetic stimulation on the autonomic nervous system and the cardiac rhythm. ScientificWorldJournal. 2014;2014:349718. doi: 10.1155/2014/349718. Epub 2014 Jul 17. PMID 25136660
- [Background] Zarate CA Jr, Mathews DC, Furey ML. Human biomarkers of rapid antidepressant effects. Biol Psychiatry. 2013 Jun 15;73(12):1142-55. doi: 10.1016/j.biopsych.2012.11.031. Epub 2013 Jan 29. PMID 23374639
- [Background] Niciu MJ, Mathews DC, Nugent AC, Ionescu DF, Furey ML, Richards EM, Machado-Vieira R, Zarate CA Jr. Developing biomarkers in mood disorders research through the use of rapid-acting antidepressants. Depress Anxiety. 2014 Apr;31(4):297-307. doi: 10.1002/da.22224. Epub 2013 Dec 18. PMID 24353110
- [Background] Pinna M, Manchia M, Oppo R, Scano F, Pillai G, Loche AP, Salis P, Minnai GP. Clinical and biological predictors of response to electroconvulsive therapy (ECT): a review. Neurosci Lett. 2018 Mar 16;669:32-42. doi: 10.1016/j.neulet.2016.10.047. Epub 2016 Oct 25. PMID 27793702
- [Background] Kerwin LJ, Keller CJ, Wu W, Narayan M, Etkin A. Test-retest reliability of transcranial magnetic stimulation EEG evoked potentials. Brain Stimul. 2018 May-Jun;11(3):536-544. doi: 10.1016/j.brs.2017.12.010. Epub 2017 Dec 29. PMID 29342443
- [Background] Minelli A, Abate M, Zampieri E, Gainelli G, Trabucchi L, Segala M, Sartori R, Gennarelli M, Conca A, Bortolomasi M. Seizure Adequacy Markers and the Prediction of Electroconvulsive Therapy Response. J ECT. 2016 Jun;32(2):88-92. doi: 10.1097/YCT.0000000000000274. PMID 26397151
- [Background] Smith M, Dietrich BJ, Bai EW, Bockholt HJ. Vocal pattern detection of depression among older adults. Int J Ment Health Nurs. 2020 Jun;29(3):440-449. doi: 10.1111/inm.12678. Epub 2019 Dec 6. PMID 31811697